CLINICAL TRIAL: NCT07099846
Title: The Use of Hyaluronic Acid and Polynucleotides in Ridge Preservation Sites Rehabilitated With a Complete Full Digital Workflow
Brief Title: Hyaluronic Acid and Polynucleotides in Ridge Preservation
Acronym: P-005
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-005
Record Dates: First submitted 2025-05-08; First posted 2025-08-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Socket Preservation; Implant-supported Single Crowns; Hyaluronic Acid; CAD-CAM
Keywords: alveolar ridge preservation; hyaluronic acid; polynucleotides; digital workflow; CAD-CAM; Implant rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous post extraction healing (No Intervention): The control group will not receive any biomaterial in the post extraction socket
- Alveolar ridge preservation (Experimental): In the group assigned to receive socket preservation, particulate deproteinizied bovine bone mineral (Bio-oss, Geistlich biomaterials) mixed with a gel containing hyaluronic acid and polynucleotides (Regenfast, Mastelli) will be placed in the socket without overfilling it and the socket will be sealed with a porcine collagen matrix (Mucograft seal, Geistlich), Any remaining PNHA gel will be placed at the entrance of the socket and on the surrounding gingival tissue
  Interventions: Device: regeneration of post extraction socket with biomaterials

INTERVENTIONS:
Device: regeneration of post extraction socket with biomaterials — after tooth extraction, in the test group we will place a demineralised bovine bone graft mixed with a gel containing hyaluronic acid and polynucleotide and we will cover the entrance of the socket with a collagen matrix
  Other Names: alveolar ridge preservation; socket preservation
  Arms: Alveolar ridge preservation

SUMMARY:
The aim of this study is to test the use of a bovine-derived bone graft combined with a polynucleotides-rich hyaluronic acid (PNHA) gel for the preservation of the bone after a tooth extraction (alveolar ridge preservation) and to test the performance of a fully-digital workflow to rehabilitate the site with a dental implant. 40 patients in need for a single tooth extraction will be recruited at Centro di Odontoiatria, Università di Parma and they will be randomly assigned to 2 groups: extraction and spontaneous healing or extraction and regeneration of the site with a bovine-derived bone graft combined with a PNHA gel. At 4 months after extraction an implant will be placed in the extraction site, which will be rehabilitated with a fully-digital workflow and patients will be followed up at up to 12 months post rehabilitation. Two 3D x-rays with a small field of view will be performed immediately after extraction and at 4 months post extraction to plan implant placement. These images will also be used to assess changes in the dimension of the post extraction bone (primary outcome). As part of the study different questionnaires will be administered to assess quality of life and perception of the therapy and the wound exudate in the area of the extraction will be collected non invasively with a collagen sponge to assess the expression of different proteins during the early healing days. On the day of implant placement a sample of bone tissue will also be collected as part of the bone drilling and histologically analysed.

DETAILED DESCRIPTION:
This is a single-centre, double-blind RCT involving 40 patients in need for a single tooth extraction to be replaced with a dental implant. The study consists of 11 visits, over a minimum period of 20 months. Participants will be recruited at Centro di Odontoiatria, at Università di Parma amongst patients routinely seen in new patient clinics and follow-up clinics. After atraumatic tooth extraction, participants will be randomly allocated to one of the following treatment groups: - DBBM (Bio-oss, Geistlich) mixed with a PNHA gel (Regenfast, Mastelli) and socket sealed with a porcine collagen matrix (Mucograft seal, Geistlich) (Test); - Unassisted socket healing (Control). Patient post-operative discomfort will be assessed with a visual analogue scale (VAS) and through clinician-reported post-operative oedema/swelling. Clinical evaluation of socket healing and recording of soft tissue healing index of Landry will also be performed during the early post-extraction days. With the help of a sterilecollagen sponge, wound exudate will be collected at 3, 7 and 14 days post extraction. A CBCT with a small field of view (e.g. 5X8 cm) will be taken to assess the post-extraction socket dimensions and after 4 months to plan implant placement. The CBCT scan will be processed with its embedded segmentation function to remove scattering defects and obtain the maximal possible quality.

Changes in alveolar ridge width from the extraction until 4 months post extraction between the 2 groups will be assessed with a dedicated software (e.g. SMOP) (primary outcome).

On the day of implant placement, a bone core biopsy will be collected from the drilling site. Undecalcified histology analysis will be done, and qualitative histology will be performed by a blind examiner, who will assess the level of maturation of the tissue in the two groups. Moreover, histomorphometric measurements will be recorded and presented descriptively, including amount of mineralized bone, as well as other standard parameters, such as %graft particles (test group only) and % of immature woven bone. A fully digital workflow will be followed to rehabilitate the patients, which will be followed up at up to 12 months post implant loading.

ELIGIBILITY:
Inclusion Criteria:

* ≥25-year-old males and females;
* good systemic health (self-assessment);
* presence of an unrestorable/hopeless tooth with periodontal attachment and buccal bone preserved at least for 2/3rd of the root and not associated with acute periapical pathology;
* full mouth bleeding and plaque scores ≤ 25%

Exclusion Criteria:

* uncontrolled or untreated periodontal disease;
* history of local (head and neck) radiation therapy in the past 5 years;
* acute endodontic lesion in the test tooth or in the neighbouring areas to the extraction procedure (sites with presence of an asymptomatic chronic lesion are eligible);
* medical history that includes uncontrolled diabetes or hepatic or renal disease, or other serious medical conditions that can impact on bone metabolism (e.g. rheumatoid arthritis, osteoporosis) or transmittable diseases (e.g. HIV-related disease);
* history of alcohol or drug abuse;
* smokers of ≥10 cigarettes a day;
* self-reported pregnancy or lactation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in alveolar ridge width at 4 months post extraction between study groups | 4 months after tooth extraction (visit 6)
  This is a superiority outcome evaluating horizontal ridge width changes at four months post-extraction between test and contro group with the help of a CBCT scan.

SECONDARY OUTCOMES:
quality of newly formed bone | 4 months post extraction (visit 6)
  to qualitatively assess socket healing and the maturity of the newly formed bone when DBBM combined with a PNHA and covered by a collagen matrix is employed for alveolar ridge preservation as compared to unassisted healing . A bone core biopsy will be taken at 4 months in both groups and the percentage of connective tissue, woven bone and mineralised bone calculated
3D volume changes | 4 months post extraction (visit 6)
  to assess 3D volume changes in soft and hard tissues at 4 and 12 months post extraction (this will be performed after digitally superimposing DICOM and STL files and in a selected region of interest) in the test and control groups
changes in protein expression | 3, 7 and 14 days post extraction (Visit 3, 4, 5)
  to assess and compare the expression of proteins and signalling pathways in the wound exudate at early healing stages. This will be done through full proteomic analysis via mass spectrometry of the wound exudate
Profilometric changes | 3, 7, 14 days and at 4 months post extraction (visit 3, 4, 5)
  to assess profilometric changes in the alveolar ridge via superimposition of intra oral scans of test and control groups
Change in post operative discomfort | 3, 7 and 14 days after extraction (visit 3, 4, 5)
  to assess changes in patient post-operative discomfort, interference with daily activities and oedema and clinician-reported post-operative oedema/swelling via visual analogue scale (VAS) scale going from 0 (no effect) to 10 (maximum negative effect)
Change in Landry healing index | 3, 7 and 14 days after extraction (Visit 3, 4, 5)
  to assess changes in soft tissue healing index of Landry (qualitative index measured with a visual scale) in the test and control groups
Changes in keratinized tissue | 4 months post extraction (Visit 6) and at study termination 12 months post loading (Visit 10);
  to assess changes in keratinized tissue (KT) height (measured in mm) in the area of the extraction (with the help of a periodontal probe) in the test and control groups
Qualitative assessment of post-operative need for medications | Starting after extraction (visit 2) and until 14 days post extraction (Visit 3, 4, 5)
  To record self-reported dosage and type of medications taken by the patients to control post operative pain in the test and control groups
Possibility to prosthetically place an implant | implant placement (Visit 7 - within 5 months from tooth extraction)
  To qualitatively describe the ability or not to place the implant in a prosthetically guided implant position with the endosteal portion of the implant completely in bone with more than 1-1.5 mm thickness on the buccal and oral aspect (Tonetti et al., 2023) (i.e. need for regeneration) at implant placement
Peri-implant radiographic bone level changes | at implant loading (visit 9 - within 5 months from implant placement) and at the end of the study (12 months post loading - visit 10)
  To assess on peri-apical x-rays the changes in peri-implant bone levels (distance between bone crest and implant shoulder) in the 2 groups
Participants' satisfaction with treatment | at the end of the study, 12 months post loading (Visit 10)
  To qualitatively report participants' satisfaction via visual analogue scale (VAS) scale going from 0 (worse) to 10 (maximum positive effect)
Implant torque | Implant placement (visit 7 - within 5 months from tooth extraction)
  To qualitatively report implant torque, which is assessed with a torque wrench after surgically placing the implant and is measured in N/cm

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro di Odontoiatria, Dipartimento di Medicina e Chirurgia, Università di Parma, Parma
  - Centro di Odontoiatria, Parma

IPD SHARING:
Plan to Share IPD: No
All patients' data held will be coded and pseudo-anonymised with an alphanumerical code that will be kept separately from the personal data as name, surname, date and place of birth and sex and stored in a locked cabinet in the PI's office.
  The only people within the Centro di Odontoiatria who will have access to information that identifies the patients will be people who need to contact them about the research study, and make sure that relevant information about the study is recorded for their care, and to oversee the quality of the study or audit the data collection process. The people who analyse the information will not be able to identify patients and will not be able to find out their name or contact details.

REFERENCES:
- [Background] Guizzardi S, Galli C, Govoni P, Boratto R, Cattarini G, Martini D, Belletti S, Scandroglio R. Polydeoxyribonucleotide (PDRN) promotes human osteoblast proliferation: a new proposal for bone tissue repair. Life Sci. 2003 Aug 29;73(15):1973-83. doi: 10.1016/s0024-3205(03)00547-2. PMID 12899922
- [Background] Colangelo MT, Govoni P, Belletti S, Squadrito F, Guizzardi S, Galli C. Polynucleotide biogel enhances tissue repair, matrix deposition and organization. J Biol Regul Homeost Agents. 2021 Jan-Feb;35(1):355-362. doi: 10.23812/20-320-L. No abstract available. PMID 33480222
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987